CLINICAL TRIAL: NCT02922764
Title: A Phase 1 Study of RGX-104, a Small Molecule LXR Agonist, as a Single Agent and as Combination Therapy in Patients With Advanced Solid Malignancies and Expansion in Select Malignancies
Brief Title: A Study of RGX-104 in Patients With Advanced Lung & Endometrial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inspirna, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGX-104-001
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Cancer; Endometrial Cancer Recurrent; Lung Cancer Recurrent; Lung Cancer; Non-small Cell Lung Cancer Metastatic; Non-small Cell Carcinoma
Keywords: Solid malignancy; Solid tumor; Non-small cell lung cancer; NSCLC; LXR; ApoE; Small cell lung cancer; SCLC; Endometrial; Endometrial Cancer; Malignant Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Neoplasms | interventions — Ipilimumab; Docetaxel; pembrolizumab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Recurrent NSCLC (2nd/3rd Line Lung Cancer). Expansion (Experimental): RGX-104 in combination docetaxel
  RGX104 120 mg BID (5day on/2days off)
  Interventions: Drug: RGX-104; Drug: Docetaxel
- Newly dignosed NSCLC Cohort Expansion (Experimental): RGX104 + pembrolizumab + carboplatin/pemetrexed
  RGX104 120 mg BID (5day on/2days off)
  Interventions: Drug: RGX-104; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed
- Recurrent/Relapsed Small Cell Lung Cancer (SCLC) Expansion (Experimental): RGX-104 + docetaxel
  RGX104 120 mg BID (5day on/2days off)
  Interventions: Drug: Docetaxel
- Recurrent/Relapsed Endometrial Cancer Expansion (Experimental): RGX-104 combined with ipilimumab
  RGX104 120 mg BID (5day on/2days off)
  Interventions: Drug: RGX-104; Drug: Ipilimumab

INTERVENTIONS:
Drug: RGX-104
  Arms: Newly dignosed NSCLC Cohort Expansion; Recurrent NSCLC (2nd/3rd Line Lung Cancer). Expansion; Recurrent/Relapsed Endometrial Cancer Expansion
Drug: Ipilimumab
  Arms: Recurrent/Relapsed Endometrial Cancer Expansion
Drug: Docetaxel
  Arms: Recurrent NSCLC (2nd/3rd Line Lung Cancer). Expansion; Recurrent/Relapsed Small Cell Lung Cancer (SCLC) Expansion
Drug: Pembrolizumab
  Arms: Newly dignosed NSCLC Cohort Expansion
Drug: Carboplatin
  Arms: Newly dignosed NSCLC Cohort Expansion
Drug: Pemetrexed
  Arms: Newly dignosed NSCLC Cohort Expansion

SUMMARY:
Study RGX-104-001 is a Phase 1, first-in-human, dose escalation and expansion study of RGX-104, an oral small molecule targeting the liver X receptor (LXR), as a single agent and in combination with nivolumab, ipilimumab, docetaxel, or pembrolizumab plus carboplatin/pemetrexed.

DETAILED DESCRIPTION:
RGX-104 activates LXR, resulting in depletion of both myeloid-derived suppressor cells (MDSCs) as well as tumor blood vessels. MDSCs block the ability of T-cells and other cells of the immune system from attacking tumors.

During the dose escalation stage, multiple doses and schedules of orally administered RGX-104 with or without nivolumab, ipilimumab, docetaxel, or pembrolizumab plus carboplatin/pemetrexed (single agent or combination therapy) will be evaluated in patients with advanced solid tumors and lymphoma (i.e., locally advanced and unresectable, or metastatic) who have had progressive disease (PD) on available standard systemic therapies or for which there are no standard systemic therapies of relevant impact. Dose escalation in combination with pembrolizumab plus carboplatin/pemetrexed will be restricted to patients with non-small cell lung cancer (NSCLC).

In the expansion stage of the study, additional patients with endometrial cancer, epithelial ovarian carcinoma (EOC), NSCLC, or small cell lung cancer (SCLC)/high-grade neuroendocrine tumors (HG-NET) will be treated at the MTD (or maximum tested dose if no MTD is identified, or dose below the MTD if there is evidence suggesting a more favorable risk/benefit profile). This stage will provide further characterization of the safety, efficacy, PK, and pharmacodynamics, including biomarkers of immunologic activity and LXR target activation, of RGX-104 as a single agent (EOC), in combination with docetaxel (SCLC/HG-NET), and and in combination with pembrolizumab plus carboplatin/pemetrexed (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have histologic or cytologic evidence of a malignant solid tumor or lymphoma (any histology) and must have advanced disease, defined as cancer that is either metastatic or locally advanced and unresectable (and for which additional radiation therapy or other locoregional therapies are not considered feasible).
2. With the exception of dose escalation with pembrolizumab plus carboplatin/pemetrexed, patients enrolled in the dose escalation stages must have disease that is resistant to or relapsed following available standard systemic therapy, or for which there is no standard systemic therapy or reasonable therapy in the physician's judgment likely to result in clinical benefit or if such therapy has been refused by the patient. Documentation of the reason must be provided for patients who have not received a standard therapy likely to result in clinical benefit.
3. Patients enrolled in the expansion stages: Optional tumor biopsy may be obtained during the screening period and toward the beginning of Cycle 2 or at the time of PD, if earlier. If a biopsy is deemed by the investigator to not be in the patient's best interest, prior approval must be obtained from the Medical Monitor to waive this requirement.
4. The patient must have disease that is measurable by standard imaging techniques per RECIST or immune-related response criteria (irRC; all tumor types except lymphoma) or International Working Group (IWG) revised response criteria for malignant lymphoma (lymphoma only). For patients with prior radiation therapy, measurable lesions must be outside of any prior radiation field(s), unless disease progression has been documented at that disease site subsequent to radiation.
5. The patient is ≥18 years old.
6. The patient has an ECOG PS of ≤1.
7. The patient has adequate baseline organ function, as demonstrated by the following:

   * Serum creatinine ≤1.5 × institutional upper limit of normal (ULN) or calculated creatinine clearance >30 mL/min (>45 ml/min for patients receiving carboplatin/pemetrexed).
   * Serum albumin ≥2.5 g/dl;
   * Bilirubin ≤1.5 × institutional ULN.
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × institutional ULN. Patients enrolled in an expansion stage may have ALT and AST < 5 × institutional ULN if the patient has hepatic metastases;
   * For patients not taking warfarin or other oral anticoagulants: international normalized ratio (INR) ≤1.5 or prothrombin time (PT) ≤1.5 × ULN; and either partial thromboplastin time or activated partial thromboplastin time (PTT or aPTT) ≤1.5 × ULN. Patients taking warfarin should be on a stable dose that results in a stable INR <3.5. Among patients receiving other oral anticoagulant therapy, PT or aPTT must be within the intended therapeutic range of the anticoagulant.
8. The patient has adequate baseline hematologic function, as demonstrated by the following:

   * Absolute neutrophil count (ANC) ≥1.5×109/L;
   * Hemoglobin ≥8 g/dL and no red blood cell (RBC) transfusions during the prior 14 days;
   * Platelet count ≥100×109/L and no platelet transfusions during the prior 14 days.
9. The patient has a normal left ventricular ejection fraction (LVEF) per institutional criteria as determined by either echocardiography (ECHO) or multigated acquisition (MUGA) scanning.
10. If the patient is a woman of child-bearing potential (WOCBP), she has had a negative serum or urine pregnancy test within 2 weeks prior to treatment.
11. The patient (men and WOCBP) agrees to use acceptable contraceptive methods for the duration of time on the study, and continue to use acceptable contraceptive methods for 1 month after the last dose of study therapy. Patients receiving combination therapy must agree to use acceptable contraceptive methods for the duration of time on the study and continue to use acceptable contraceptive methods for 6 months after the last dose of study therapy.
12. The patient has signed informed consent prior to initiation of any study-specific procedures or treatment.
13. The patient is able to adhere to the study visit schedule and other protocol requirements, including follow-up for survival assessment.
14. Tumor tissue (a minimum of 10 and up to 15 unstained slides, or paraffin block, ideally from the patient's most recent biopsy, must be made available prior to the first dose of study therapy.
15. For patients with endometrial cancer enrolled in the ipilimumab combination expansion stage:

    * The patient has Stage III, Stage IV, or recurrent, histologically-confirmed endometrial carcinoma with disease that is measurable per RECIST 1.1.
    * The patient may have received up to THREE lines of prior therapy:

    Prior systemic platinum-based adjuvant and/or neoadjuvant chemotherapy counts as one prior line of therapy.

    A prior systemic therapy for advanced or recurrent disease counts as one prior line of therapy (if not given in the adjuvant or neoadjuvant setting).

    A prior checkpoint inhibitor therapy (anti PD-1/PD-L1) with or without an angiogenesis inhibitor counts as one prior line of therapy.

    Prior hormone and radiation therapy is not counted as prior therapies. The patient has either archival tumor tissue sample available (preferable) or in the absence has documented determination of mismatch repair (MMR) status.
    * The patient may not have received treatment with immune checkpoint inhibitors (e.g., products that target PD-L1, PD-1, or CTLA-4).
    * The patient must not have required a paracentesis within the preceding 4 weeks nor be projected to require a paracentesis within the next 8 weeks.
16. For patients with NSCLC enrolled in the pembrolizumab plus carboplatin/pemetrexed combination dose escalation or expansion stages:

    * The patient must have histologic or cytologic evidence of newly-diagnosed non-squamous, NSCLC that is advanced disease, defined as cancer that is either metastatic (Stage 4) or locally advanced (Stage 3B) and unresectable.
    * The patient has confirmation that epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK)-directed therapy is not indicated.
    * The patient has not received prior systemic treatment for their advanced/metastatic disease.
    * For patients in the expansion stage only: the patient's tumor block must demonstrate PD-L1 expression TPS <1% as determined with a validated assay.
    * The patient must have adequate organ function and performance status eligible for treatment with a platinum-based regimen and checkpoint inhibitor.

Exclusion Criteria:

1. The patient has persistent clinically significant toxicities (Grade ≥2) from previous anticancer therapy (excluding Grade 2 chemotherapy-related neuropathy and alopecia which are permitted). Prior toxicities that resulted in laboratory abnormalities should have resolved to Grade ≤1, unless a higher-grade abnormality is allowed by the inclusion criteria. If medical therapy is required for the treatment of a laboratory abnormality, the dose and laboratory value(s) should be stable.
2. If considered for combination therapy with nivolumab or ipilimumab, the patient has:

   * Uncontrolled clinically significant pulmonary disease.
   * A history of any grade immune-related ocular event.
   * A history of Grade ≥3 immune-related adverse event regardless of offending agent.
   * Active autoimmune disease that required systemic treatment in the past. Patients who have not required systemic treatment for at least two years may be enrolled if permission is provided after discussion with the Medical Monitor (replacement therapy, e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, is not considered a form of systemic treatment, and is allowed).
   * Evidence of active noninfectious pneumonitis or history of interstitial lung disease.
   * A risk of reactivation of hepatitis B or C.
   * Previously received an immune therapy that was discontinued due to immune-related AEs, regardless of grade.
   * Uncontrolled endocrine disorder. Patients who are on endocrine replacement therapy must be on a stable dose.
3. The patient has received treatment with chemotherapy, external-beam radiation, or other systemic anticancer therapy within 14 days prior to study therapy administration (42 days for prior nitrosourea or mitomycin-C; patients with advanced prostate cancer who are receiving luteinizing hormone releasing hormone (LHRH) agonists are permitted onto the study and should continue use of these agents during study treatment).
4. The patient has received treatment with an investigational systemic anticancer agent within 14 days prior to study therapy administration.
5. The patient has previously received treatment with RGX-104 or another investigational agent that is a known LXR agonist.
6. The patient has an additional active malignancy that may confound the assessment of the study endpoints. Patients with a past cancer history with substantial potential for recurrence must be discussed with the Medical Monitor before study entry. Patients with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including transitional cell carcinoma, cervical intraepithelial neoplasia, and melanoma in situ), organ-confined prostate cancer with no evidence of progressive disease.
7. The patient has clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association Class 3 or 4 heart failure (see Appendix 1), uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
8. The patient has uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the patient at significant risk for pulmonary complications during the study.
9. The patient has known active or suspected brain or leptomeningeal metastases. Central Nervous System (CNS) imaging is not required prior to study entry unless there is a clinical suspicion of CNS involvement. Patients with stable, treated brain metastases are eligible provided there is no evidence of CNS disease growth on imaging for at least 8 weeks following radiation therapy or other locoregional ablative therapy to the CNS.
10. The patient has a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to study therapy administration. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
11. The patient has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection requiring therapy, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements.
12. The patient is pregnant or breast feeding.
13. The patient has known positive status for human immunodeficiency virus or active or chronic Hepatitis B or Hepatitis C.
14. The patient is oxygen-dependent.
15. The patient has a history of pancreatitis.
16. The patient has Grade ≥2 hypercholesterolemia (total cholesterol >300 mg/dL or >7.75 mmol/L) and/or hypertriglyceridemia (triglyceride >300 mg/dL or >3.42 mmol/L) in the fasting state.
17. QTcF >450 msec (males) or >470 msec (females).
18. The patient has a physical abnormality or medical condition that limits swallowing multiple pills, or has a history of non-adherence to oral therapies.
19. The patient requires statin (e.g., rosuvastatin, atorvastatin, etc.) therapy. If the patient is taking a statin but discontinuation is considered appropriate, the statin must be discontinued at least 5 days prior to starting study therapy.
20. The patient requires treatment with a medication that is a strong inhibitor of CYP3A4 (boceprevir, clarithromycin, conivaptan, grapefruit juice, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, or voriconazole).
21. For the docetaxel escalation stage, patients with NSCLC with alkaline phosphatase > 2.5 × institutional ULN and AST or ALT > 1.5 × institutional ULN.
22. For patients with NSCLC enrolled in the pembrolizumab plus carboplatin/pemetrexed combination dose escalation or expansion stages:

    * The patient received radiation therapy to the lung that is >30 Gray (Gy) within 6 months of the first dose of study medication
    * The patient completed palliative radiotherapy ≤7 days of the first dose of study medication
    * The patient has received live-virus vaccination ≤30 days of planned start of study medication
    * The patient has clinically active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, peritoneal carcinomatosis
    * The patient is expected to require any other form of antineoplastic therapy while on study.
    * The patient has known hypersensitivity to another monoclonal antibody (mAb)
    * The patient has known sensitivity to any component of carboplatin or pemetrexed
    * The patient is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose ≤1.3 g per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam)
    * The patient is unable or unwilling to take folic acid or vitamin B12 supplementation
23. The patient has clinical or laboratory evidence of a paraneoplastic syndrome.
24. The patient has experienced weight loss of >10% of their body weight over the preceding 3 months.
25. The patient has any medical condition which, in the opinion of the Investigator, places the patient at an unacceptably high risk for toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD), or the maximum tested dose at which multiple DLTs are not observed, of RGX-104 as a single agent, and separately, in combination with nivolumab, ipilimumab, docetaxel, or pembrolizumab plus carboplatin/pemetrexed. | 6 months
Overall response rate associated with RGX-104 treatment as a single agent, and separately, in combination with docetaxel or pembrolizumab plus carboplatin/pemetrexed. | 24 months
Progression-free survival associated with RGX-104 treatment as a single agent, and separately, in combination with docetaxel or pembrolizumab plus carboplatin/pemetrexed. | 24 months
Number of participants with treatment-emergent adverse events associated with RGX-104 treatment as a single agent, and separately, in combination with nivolumab, ipilimumab, docetaxel, or pembrolizumab plus carboplatin/pemetrexed. | 24 months

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Plasma Concentration (Cmax) of RGX-104. | 24 months
Pharmacokinetics: Area Under the Curve (AUC) of RGX-104. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wasserman, MD, Study Director — Inspirna, Inc.
Locations (21):
- United States (21):
  - Arizona Oncology, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Sarah Cannon Research Institute, Denver, Colorado
  - Florida Cancer Specialist, Lake Mary, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maryland Oncology, Columbia, Maryland
  - Regions Hospital, Saint Paul, Minnesota
  - Dartmouth Hitchcock Medical, Lebanon, New Hampshire
  - CINJ, New Brunswick, New Jersey
  - Quantum Santa Fe, Santa Fe, New Mexico
  - Columbia University Medical Center, New York, New York
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Virginia Cancer Specialists, PC, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No